CLINICAL TRIAL: NCT01691092
Title: PET Imaging of mGluR5 With Drug Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1111009365
Record Dates: First submitted 2012-09-19; First posted 2012-09-24 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Major Depressive Disorder; Post-Traumatic Stress Disorder (PTSD)
Keywords: Depression; Ketamine; PET; PTSD
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Depression | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketamine (Experimental): All subjects will receive ketamine
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — All subjects will receive ketamine to induce glutamate release in the brain
  Other Names: ketamine IV

SUMMARY:
This study is designed to look at that involvement of a process in the brain called the glutamate system in depression. Participants will undergo a screening session, up to two functional Magnetic Resonance Imaging (fMRI) scans, and up to three Positron Emission Tomography (PET) scans, as well as cognitive testing at each scan session. For one of the PET scans, a drug (either ketamine or n-acetyl cysteine) will be administered.

Hypothesis 1: The investigators hypothesize administration of ketamine or n-acetylcysteine (NAC) will lead to a decrease in mGluR5.

Hypothesis 2: The investigators hypothesize an improvement in memory and attentional skills after drug challenge.

Hypothesis 3: The investigators hypothesize an increase in mGluR5 availability and change in MRI measures post drug challenge as compared to baseline, signifying synaptogenesis.

Hypothesis 4: We expect there should not be a significant difference in reduction in mGluR5 availability due to differences in ABP688 radiotracer infusion.

DETAILED DESCRIPTION:
Aim 1: To determine the acute effect of medication-induced glutamate release on mGluR5 availability in human subjects. Hypothesis 1: We hypothesize administration of ketamine or n-acetylcysteine (NAC) will lead to a decrease in mGluR5 availability.

Aim 2: To determine if glutamate release via administration of ketamine or NAC has pro cognitive benefits.

Hypothesis 2: We hypothesize an improvement in memory and attentional skills after drug challenge.

Aim 3: To determine if there is synaptogenesis detectable by PET and MRI post ketamine or NAC within a week of drug challenge (at the time of greatest antidepressant response). Hypothesis 3: We hypothesize an increase in mGluR5 availability and change in MRI measures, post drug challenge as compared to baseline, signifying synaptogenesis.

Aim 4: To determine if there is a difference in reduction of mGluR5 availability after ketamine administration when radiotracer is administered bolus as compared to bolus to constant infusion in the same subjects (ABP688 radiotracer only).

Hypothesis 4: We expect there should not be a significant difference in reduction in mGluR5 availability due to differences in ABP688 radiotracer infusion.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* English speaking
* No other Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (DSM-IV) diagnosis present, besides required as below.

Inclusion criteria for depressed subjects

* clinical diagnosis of a current or past depressive episode
* medication free for at least 2 weeks
* Score >16 on Hamilton Depression Rating Scale (HDRS) if currently depressed or <11 if not currently depressed
* treatment or non-treatment seeking who understand that this study is for research purposes only

Inclusion criteria for healthy controls

* no current, or history of, any DSM-IV diagnosis
* no first-degree relative with history of psychotic, mood, or anxiety disorder

Inclusion criteria for PTSD subjects

* current Post-Traumatic Stress Disorder, as determined by the Structured Clinical Interview for DSM-IV-Text Revision (TR) (SCID) patient research edition
* Clinician Administered PTSD Scale for DSM-IV-TR (CAPS) score of 50 or higher

Inclusion criteria for trauma control subjects

-history of trauma (meeting the criterion A of PTSD but not a full diagnosis of PTSD)

Exclusion Criteria:

* Current or past significant medical, neurological, or metabolic disorder or loss of consciousness for 5 minutes or more
* active, significant suicidal ideation
* implanted metallic devices or any Magnetic Resonance (MR) contraindications
* women who are pregnant or breastfeeding
* met DSM-IV criteria for alcohol/illicit substance dependence in their life-time or met alcohol/illicit substance abuse within past year
* history of prior radiation exposure for research purposes within the past year such that participation in this study would place them over FDA limits for annual radiation exposure. This guideline is an effective dose of 5 rem received per year
* blood donation within eight weeks of the start of the study
* radiation exposure at work that precludes study participation
* blood pressure >140/80

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irina Esterlis, PhD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Connecticut Mental Health Center, New Haven, Connecticut
  - Yale University Magnetic Resonance Research Center (MRRC), New Haven, Connecticut
  - Yale University PET Center, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine
Started | 79
Completed | 38
Not Completed | 41
Not completed — Lost to Follow-up | 10
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 3
Not completed — non-compliance | 3
Not completed — used for different study | 2
Not completed — screen fail | 19

BASELINE CHARACTERISTICS:
Population: reason for discrepancy: some subjects completed baseline scan but did not continue with ketamine administration and subsequent scans.
Arm/Group | Ketamine
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.07143 (12.12615)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 14
diagnosis [Count of Participants; unit: Participants]
  Healthy Control (HC) | 20
  Major Depressive Disorder (MDD) | 14
  Post-Traumatic Stress Disorder (PTSD) | 4
  Comorbid MDD & PTSD | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Glutamate Levels at Baseline and After Ketamine Administration as Confirmed by Positron Emission Tomography (PET) Imaging
Description: PET imaging obtained in healthy and Major Depressive Disorder (MDD) subjects. Glutamate levels determined by radiotracer uptake in PET images.
Time Frame: 1st scan: 90 minute baseline scan; 2nd scan: 90 minutes, ketamine administration at start of scan; scan 3: 90 minute scan 24 hours post ketamine
Population: 13 healthy (6 males, 7 females) and 14 MDD non-smokers (4 males, 10 females) Mean age: 33.5 ± 13.2 yrs reasons for discrepancy (participant flow module): some data was not able to be analyzed due to elevated metabolites; some subject did not tolerate ketamine and had to be pulled out of scanner so we could not obtain data.
Measure: Mean (Standard Deviation); unit: percentage reduction
Arm/Group | Ketamine
Number analyzed (Participants) | 27
percentage reduction
  HC % reduction from baseline immediately post ket | 19 (22)
  MDD % reduction from baseline immediately post ket | 14 (9)
  HC % reduction from baseline 24 hrs post ket | 31 (30)
  MDD % reduction from baseline 24 hrs post ket | 14 (13)

ADVERSE EVENTS:
Time Frame: 4 years
Description: Standard assessments and regular observations are used to determine whether or not certain adverse events have occurred.
Arm/Group | Ketamine
Serious Adverse Events (participants affected / at risk) | 1/38
Other Adverse Events (participants affected / at risk) | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=38)
post-ketamine non-responsiveness (General disorders) | 1 (1) — Post-ketamine subject was non-responsive to questions- did not respond to verbal arousal. Subject was clinically stable. Sent to ER where it was believed the experience was dissociative event due to ketamine.

LIMITATIONS AND CAVEATS:
Study lacks placebo control group Hemodynamic effects of ketamine may alter tracer delivery and washout Study lacks long-term follow up Only non-smokers studied Ketamine dose administered is higher than typical dose used for clinical purposes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No